CLINICAL TRIAL: NCT03052738
Title: Medical Marijuana in the Pediatric Central Nervous System Tumor Population
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0404.cc
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Central Nervous System Tumor; Brain Tumor; Spinal Tumor
Keywords: central nervous system (brain or spinal) tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Spinal Cord Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study proposes to do a prospective observational cohort study evaluating the quality of life (QOL) of children with Central Nervous System (CNS) tumors and their families who choose to self-medicate with marijuana-derived products while undergoing treatment at Children's Hospital Colorado (CHCO).

DETAILED DESCRIPTION:
Children's Hospital Colorado (CHCO) Center for Cancer and Blood Disorders (CCBD) is a national leader in pediatric cancer therapy. The CHCO Neuro-Oncology program treats more that 90% of Coloradan children with Central Nervous System (CNS) tumors and a large percentage of children with CNS tumors from the surrounding five states. Due to advances in therapy, approximately two-thirds of children with CNS tumors treated at CHCO will be cured. Although medical marijuana has been legal for more than a decade in Colorado, the publicity around the more recent legalization for general adult use, increasing literature, and anecdotal reports of patients with terminal CNS tumors cured with medical marijuana, have prompted a recent increase in interest of current CHCO patients and their families. There has been an influx of pediatric cancer patients and their families moving to Colorado to obtain these marijuana-based products to self-medicate.

The Investigators will administer PedsQLTM questionnaires and diaries to gather data regarding use practices, method of delivery, strain used, dosing and frequency, and family financial impact on all enrolled patients. The Investigators will also collect peripheral blood samples to evaluate for evidence of immuno-modulation by cannabinoids in patients who may already be immunocompromised and to assess blood cannabinoid levels.

This study will provide novel exploratory data regarding use patterns, impact on families and resources, and potential clinical benefits and harms associated with the growing marijuana use in the pediatric neuro-oncology population. Such information may guide future children afflicted with CNS tumors and their families to make decisions about whether to pursue cannabinoid treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 2 years and < 18 years at the time of study enrollment.
2. Parents/legal guardian(s) that will be completing the questionnaires must sign consent. There are no age parameters for parent/legal guardians' participation on study.
3. Patients must have a diagnosis of central nervous system (brain or spinal) tumor
4. Patients must be ONE of the following:

   * Undergoing disease-directed therapy or disease surveillance as prescribed by the Pediatric Neuro-Oncology physicians at CHCO
   * Planning to transfer medical care to Pediatric Neuro-Oncology physicians at CHCO from outside facilities
   * Receiving palliative care services that are managed in conjunction with physicians at CHCO
5. Interest in marijuana use has been discussed by the patient or parents.
6. Patient has not used any marijuana products or synthetics in the last 14 days (a washout period of 14 days is permitted for those interested in participating on this study)

   1. An exception to this rule is if patients took their first dose within 72 hours of signing consent. These patients will be eligible for study without going through a washout period.

Exclusion Criteria:

1. Does not meet inclusion criteria
2. Use (or planned use) of synthetic marijuana products as sole cannabinoid therapy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a prospective observational cohort study evaluating the quality of life (QOL) of children with CNS tumors and their families who choose to self-medicate with marijuana-derived products while undergoing treatment at CHCO.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Overall Quality of Life | 1 year
  quality-of-life scores as assessed by the validated PedsQL™ brain tumor (PedsQL™-BT) module

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas K Foreman, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Chilsdren's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No